CLINICAL TRIAL: NCT01747772
Title: Evaluate the Utility of Shear Wave Sonoelastography as a Tool to Measure Liver Fibrosis Grade
Brief Title: Sonoelastography: Ultrasound Method to Measure Liver Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Anthony Samir, Associate Director, Ultrasound Imaging Services Assistant Radiologist, Abdominal Imaging & Intervention Massachusetts General Hospital, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2009P002791
Record Dates: First submitted 2012-10-31; First posted 2012-12-12 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Chronic Liver Disease; Non-Alcoholic Fatty Liver Disease; Hepatitis C Virus (HCV) Coinfection; Hepatitis B Virus (HBV); Drug-Induced Liver Injury
Keywords: Non-focal Liver Disease; Fibrosis; Shear Wave Sonoelastography; Metavir Liver Fibrosis Grading
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Hepatitis C; Coinfection; Hepatitis B; Chemical and Drug Induced Liver Injury; Fibrosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Biopsy specimens were assessed via Meta-analysis of Histological Data in Viral Hepatitis (METAVIR) criteria by a pathologist who was blinded to the shear-wave elastography (SWE) values.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Shear Wave Sonoelastography for Fibrosis Assessment (Experimental): Shear Wave sonoelastography (SWE) was performed in patients who were scheduled for a non-focal liver biopsy.
  Interventions: Device: Shear Wave Sonoelastography

INTERVENTIONS:
Device: Shear Wave Sonoelastography — Shear Wave sonoelastography (SWE) as an ultrasound technique to measure liver fibrosis was performed on patients scheduled for non-focal liver biopsy. Results were compared with pathological score from liver biopsy.
  Other Names: Supersonic Aixplorer

SUMMARY:
HYPOTHESIS: The investigators hypothesize that sonoelastography (SE) will provide accurate quantitative measurements that can be used to stage liver fibrosis in patients with chronic liver disease.

1. To measure liver stiffness with sonoelastography in adults with suspect diffuse liver disease who will undergo non-focal liver biopsy as part of their routine clinical care
2. To assess the sensitivity and specificity of sonoelastography for the detection and staging of liver fibrosis
3. To evaluate the effect of steatosis and inflammation on the estimation of liver fibrosis using sonoelastography

DETAILED DESCRIPTION:
BACKGROUND Chronic liver disease is an important cause of morbidity and mortality in the United States. A retrospective cohort study identified 2,353 patients with newly diagnosed chronic liver disease (63.9 cases/100,000 population). Extrapolating this incidence rate there will be approximately 150,000 patients with chronic liver disease diagnosed in gastroenterology clinics each year. Almost 20%, or an estimated 30,000 patients per year, had established cirrhosis at the time of presentation to the gastroenterologist.

Cirrhosis remains a major public health problem and disease-related complications were associated with nearly 40,000 deaths and more than 1.4 billion dollars spent on medical services in the United States. There is a great need to develop and identify methods of risk stratification and prognostication for patients with chronic liver disease. Hepatic fibrosis is the final common pathway for many different liver insults and is now known to be a dynamic process that is at least partially reversible. The diagnosis and quantification of fibrosis relies on liver biopsy, and liver biopsy is currently the gold standard for detecting and staging hepatic fibrosis. However, liver biopsy is an invasive procedure with significant risks, including hemorrhage, infection and visceral perforation. In addition, liver biopsy is a poor gold standard, because it is limited by interobserver variability in interpretation and sampling errors in 25-45% of cases.

A number of indirect markers and indices of liver fibrosis have been used in clinical practice. Noninvasive tests can be distinguished by direct vs. indirect measures of fibrosis and also classified by the modality of the test as serum vs. imaging. Biomarkers of the structural elements of fibrogenesis and the key inflammatory mediators involved in the genesis or degradation of scar tissue are often referred to as direct components. Indirect markers can reflect the accompanying alterations in hepatic function.

Fibrotic livers demonstrate increased stiffness. This property can be exploited and measured using a newly developed ultrasound technology named Ultrasound Elastography (Transient Elastography (TE) or sonoelastography (SE). SE is performed by insonating the patient with a low energy, low amplitude, and low frequency shear wave created by focused ultrasound or by a vibrating probe on the skin. The small tissue movements produced by the propagated wave are then measured with ultrasound. The propagated wave travels faster with increasing fibrosis: the stiffer the tissue, the faster the shear wave propagates. A pulse-echo ultrasound acquisition allows measurement of the wave velocity and the results are presented as kilopascals (kPa). Tissue elasticity is calculated as the median of 10 measurements and ranges from 2.5 to 75 kPa with normal values around 5.5 kPa (Normal liver stiffness ranges between 3.3-7.8 kPa). Hepatic stiffness can be measured within a cylinder of tissue 1 cm wide and 4 cm in length producing an estimated sampling area that is 100 times greater than a biopsy. A meta-analysis assessing the capacity of transient elastography to diagnose moderate fibrosis found pooled estimates for sensitivity and specificity of 70% and 84% respectively. The mean area under the receiver operating characteristic curve (AUROC) for the diagnosis of significant fibrosis was 0.84% with an optimal cut-off of 7.6 kPa, and the diagnostic accuracy of SE for cirrhosis had an AUROC ranging from 0.90- 0.99 (mean AUROC 0.94) and cut-off from 9.0 to 26.5 kPa. The benefits of SE are that it is inexpensive, reproducible, painless, rapid (<10 min), easy to perform, and can be used for diagnosis, prognosis and monitoring disease progression. Limitations of sonoelastography are that measurements cannot be obtained in the presence of marked obesity, ascites, or unusually narrow intercostal spaces when externally applied vibrating shear wave generators are used.

SPECIFIC AIMS

1. To evaluate liver stiffness with the diagnostic imaging method of sonoelastography among adults with suspect liver diseases.
2. To obtain estimates of the sensitivity and specificity of sonoelastography for the detection and staging of liver fibrosis.

STUDY PROCEDURES Study Visit 1: (SE or sonoelastography )

* Sonoelastography will be performed prior to standard pre-biopsy ultrasound imaging using a FDA-approved ultrasound unit. This unit will use ultrasound energy within the limits set by the FDA for diagnostic ultrasound to create a shear wave front that is progressively distorted as it traverses the tissue. Ultrafast ultrasound imaging will then be used to detect the speed of propagation of the shear wave front.
* The unit will emit no ionizing radiation and will perform ultrasound acquisition within the acoustic power and intensity limits established by the FDA for diagnostic sonography. At these energy levels there are no known bioeffects of ultrasound. Sonoelastography measurements will require approximately 15 minutes, and will be painless.
* The unit is a cart-based ultrasound system used to perform non-invasive diagnostic ultrasound studies. The system functions in a manner identical to all diagnostic ultrasound systems and transducers for the conventional modes: B-mode, Harmonic imaging, Spatial Compounding imaging and Power Doppler. Additionally, the system uses a new imaging mode based on shear wave elastography to map tissue stiffness. The elastography mode produces color-coded images of different tissues based on their elasticity. The color scale represents a quantitative assessment of tissue stiffness, thereby allowing elasticity of tissue to be quantified in units of kilopascals (kPa).
* At the conclusion of Study Visit 1, the patient will return to usual care.

Tests and Parameters:

Sonoelastography parameters:

Mean liver stiffness (elastogram) in kilopascal (kPa). SE normal values approximately 5.5 kPa (Normal liver stiffness ranges between 3.3-7.8 kPa) Significant Fibrosis (F3): = or > 7.6 kPa, Cirrhosis (F4): = or > 9.0- 26 kPa Data Collection

Data to be collected includes:

* Gender, ethnicity, age, body mass index (BMI), history of previous and current medication use, detail history of alcohol intake, comorbidities, signs and symptoms.
* Biochemical liver tests that are typically performed as part of routine clinical care (aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (APH), gamma-glutamyl transferase (GGT), tuberculosis (TB), indirect bilirubin (IB), direct bilirubin (DB), albumin, total proteins, prothrombin time (PT)).

Other laboratory data typically performed as part of routine clinical care: red blood cells (RBC), white blood cells (WBC), platelets, glucose, creatinine, lipid profile.

Any laboratory study for the diagnosis of the suspected diffuse liver disease: Viral serology, including hepatitis C virus (HCV), hepatitis B virus (HBV), ferritin, ceruloplasmin, antimitochondrial antibody (AMA), antinuclear antibody (ANA), alphafetoprotein: Sonoelastography report, and/or histological examination by a sub-specialist pathologist:

* SonoElastography

  * Normal liver stiffness ranges between 3.3-7.8 kPa, Significant Fibrosis (F3): 7.6 kPa
  * Cirrhosis (F4): 9.0- 26 kPa
* Histology (Meta-analysis of Histological Data in Viral Hepatitis [METAVIR]):

  * F0- No fibrosis, F1- Portal fibrosis without septa, F2- Portal fibrosis with rare septa, F3- Numerous septa without cirrhosis, F4 - Cirrhosis STATISTICAL ANALYSIS Descriptive statistics will be shown as mean ± standard deviation or percentages as appropriate. The patients will be divided according to fibrosis stage. The groups' binary diagnostic by different diagnostic methods will be compared with the gold standard by McNemar's Test. We will use contingency tables to analyze the correlation between sonoelastographic measurements. Factors independently correlated with liver stiffness will be assessed by multiple regression analysis. The diagnostic performance of fibrosis and/or liver stiffness will be determined in terms of sensitivity, specificity, positive and negative predictive values, diagnostic accuracy and area under receiver operating characteristics (ROC) curves. This is a pilot study and the investigators are planning to enroll 100 participants to include in this study. With 100 patients included in this study the investigators can have a > 80% power to detect a significant diagnostic power by SonoElastography with a true AUC between of 0.85 as opposed to the null with an area under the curve (AUC) of 0.62 or lower using a two-sided test with 5% type I error. In addition, multivariate linear and logistic regression models will be used to evaluate the diagnostic power of independent factors taking into account possible confounders by patient demographic and clinical characteristics. The primary outcome of interest will be fibrosis.

RISKS AND DISCOMFORTS Ultrasound Elastography: Ultrasound elastography requires the administration of ultrasound energy at levels similar to those used in diagnostic ultrasonography. There are no known bioeffects of ultrasound at these energies.

Pregnant women are excluded from this study. There are no known risks of sonoelastography to an embryo or fetus (a developing baby still in the womb). There may be risks to an embryo or fetus that are currently unknown.

POTENTIAL BENEFITS Although knowledge about liver diseases and fibrosis has increased dramatically over the last few years, much remains to be learned. The imaging strategy that will be evaluated, ultrasound sonoelastography, has the potential to reduce the number of liver biopsies performed for the diagnosis and monitoring of hepatic fibrosis. This study is expected to provide a basis for future investigation into non-invasive imaging markers of hepatic fibrosis. Any data obtained for the purposes of this study will be available to the participant's primary physicians.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18 or older)
* Men or women
* Suspected diffuse liver disease
* Consent to participate in the study

Exclusion Criteria:

* Pregnancy
* Acute illness/cognitive impairment resulting in inability to cooperate with ultrasound.
* Patients that do not consent to ultrasound or sonoelastography.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2014-02-14 (Actual); Study Completion 2014-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony E Samir, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Samir AE, Dhyani M, Vij A, Bhan AK, Halpern EF, Mendez-Navarro J, Corey KE, Chung RT. Shear-wave elastography for the estimation of liver fibrosis in chronic liver disease: determining accuracy and ideal site for measurement. Radiology. 2015 Mar;274(3):888-96. doi: 10.1148/radiol.14140839. Epub 2014 Nov 13. PMID 25393946

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients known to have or suspected of having diffuse liver disease who were scheduled for ultrasound-guided non-focal liver biopsy were eligible for the study.
Period: Overall Study
Arm/Group | Shear Wave Sonoelastography for Fibrosis Assessment
Started | 180
Analysis Population | 164 (All participants who completed the study and had adequate SWE and liver biopsy data.)
Completed | 171
Not Completed | 9
Not completed — SWE Data Not Obtainable Prior to Biopsy | 9

BASELINE CHARACTERISTICS:
Population: The analysis population included all participants who completed the study and had adequate shear-wave sonoelastography (SWE) and liver biopsy data. 16 participants were excluded: 9 discontinued and 7 had inadequate SWE or biopsy data.
Arm/Group | Shear Wave Sonoelastography for Fibrosis Assessment
Number analyzed (Participants) | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81
  Male | 83

OUTCOME MEASURES:

1. Primary Outcome: Liver Elasticity Value Measured Using Sonoelastography (SE)
Description: Liver elasticity/stiffness was assessed via SE and compared against results of liver biopsy as read by a single pathologist using the Meta-analysis of Histological Data in Viral Hepatitis (METAVIR) 5-point scale (F [Fibrosis]0=no fibrosis, F1=portal fibrosis without septa, F2=portal fibrosis with few septa, F3=numerous septa without cirrhosis, and F4=cirrhosis). Using SE, fibrosis is measured in kilopascals (kPa) with normal values equaling approximately 5.5 kPa (normal liver stiffness ranges between 3.3-7.8 kPa). Significant Fibrosis (F3): = or > 7.6 kPa, Cirrhosis (F4): = or > 9.0- 26 kPa. A higher number corresponds to an increase in stiffness and hepatic fibrosis.
Time Frame: Day 1
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: kilopascals (kPa)
Groups:
- Fibrosis 0: Participants with no fibrosis on liver biopsy evaluation.
- Fibrosis 1: Participants with portal fibrosis without septa on liver biopsy evaluation.
- Fibrosis 2: Participants with portal fibrosis with few septa on liver biopsy evaluation.
- Fibrosis 3: Participants with numerous septa without cirrhosis on liver biopsy evaluation.
- Fibrosis 4: Participants with cirrhosis on liver biopsy evaluation.
Arm/Group | Fibrosis 0 | Fibrosis 1 | Fibrosis 2 | Fibrosis 3 | Fibrosis 4
Number analyzed (Participants) | 24 | 97 | 18 | 18 | 7
kilopascals (kPa) | 7.225 [6.106 to 8.344] | 7.332 [6.903 to 7.762] | 8.548 [7.666 to 9.429] | 12.101 [8.464 to 15.738] | 10.469 [8.592 to 12.345]

ADVERSE EVENTS:
Description: Adverse events in this study were limited to those related to the performance of sonoelastography.
Arm/Group | Shear Wave Sonoelastography for Fibrosis Assessment
Serious Adverse Events (participants affected / at risk) | 0/164
Other Adverse Events (participants affected / at risk) | 0/164

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes